CLINICAL TRIAL: NCT07185815
Title: A Prospective, Dose Escalating, Open Label, Multi-center, Phase I/IIa Study to Evaluate the Pharmacokinetics, Safety, Tolerability and Efficacy of a Subcutaneous Long-Acting Injection of Cariprazine (Cariprazine Depot) in Subjects Eligible for Treatment With Oral Cariprazine.
Brief Title: Pharmacokinetics, Safety, Tolerability and Efficacy of a Subcutaneous Long-Acting Injection of Cariprazine (Cariprazine Depot) in Subjects Eligible for Treatment With Oral Cariprazine
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mapi Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Cariprazine Depot I/IIa - 001
Record Dates: First submitted 2025-08-28; First posted 2025-09-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder (MDD); Bipolar 1 Disorder; Schizophrenia
Keywords: Long acting injection; LAI; Subcutaneous; SC; Cariprazine; Cariprazine Depot
MeSH Terms: conditions — Depressive Disorder, Major; Schizophrenia | interventions — cariprazine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental)
  Interventions: Drug: Cariprazine Depot
- Cohort 2 (Experimental)
  Interventions: Drug: Cariprazine Depot
- Cohort 3 (Experimental)
  Interventions: Drug: Cariprazine Depot MTD; Drug: Oral Cariprazine 3 mg/day

INTERVENTIONS:
Drug: Cariprazine Depot — One single dose of 22 mg
  Arms: Cohort 1
Drug: Cariprazine Depot — One single dose of 44 mg
  Arms: Cohort 2
Drug: Cariprazine Depot MTD — Three monthly doses of MTD (maximum tolerated dose)
  Arms: Cohort 3
Drug: Oral Cariprazine 3 mg/day — Oral Cariprazine 3 mg/day for three months
  Arms: Cohort 3

SUMMARY:
The purpose of this study is to assess the PK, Safety, Tolerability (all cohorts) and Efficacy (cohort 3), of once-a-month long-acting SC injection of dose escalating Cariprazine Depot in subjects eligible for treatment with oral Cariprazine.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects who meet DSM-5-TR diagnostic criteria for schizophrenia, bipolar I disorder or major depressive disorder (this inclusion criterion relates to cohorts 1 and 2 only).
* Clinically stable subjects (with no evidence of deterioration and on a stable dose of oral antipsychotic or antidepressant medication(s) other than Cariprazine for at least 4 weeks, prior to screening), receiving antipsychotic/s or antidepressant/s other than oral Cariprazine and eligible for treatment with Cariprazine 3 mg/day, with CGI-S score of 0-4.
* Men and women aged 18-64 years (inclusive).
* Body mass index (BMI) 18.5-35.
* Able to sign an informed consent form.
* Adult subjects with a current diagnosis of schizophrenia, who meet DSM-5-TR diagnostic criteria for schizophrenia, naïve to or treated with antipsychotics (this inclusion criterion relates to cohort 3 only).

Key Exclusion Criteria:

* Subjects with schizophrenia with PANSS item scores of > 4 on any of the following: P4 Excitement/Hyperactivity; P6 Suspiciousness/persecution; P7 Hostility; G8 Uncooperativeness; G14 Poor impulse control.
* Subjects with schizoaffective disorder, delirium, dementia, amnestic, or other cognitive disorders or severe personality disorders.
* Use of an investigational drug, and/or participation in clinical studies with an investigational product within 3 months prior to screening.
* History or current cardiovascular or cerebrovascular disease.
* History of seizures or conditions that lower the seizure threshold.
* Use of concomitant administration of strong or moderate CYP3A4 inhibitors.
* Use of concomitant medication of strong or moderate CYP3A4 inducers is contraindicated.
* Subjects with Suicidal Thoughts and Behaviors or has a history of suicidal ideation in the past year, or made a suicide attempt in the past 5 years.
* Subjects with a history of orthostatic hypotension and/or syncope.
* Subjects clinically stable on any dose of oral Cariprazine or add-on treatment (cohorts 1-2 only).
* Subjects with CGI-S score of 5-7.
* Subjects previously treated with partial D2 agonists, aripiprazole and brexipiprazole, and suffered from clinically relevant akathisia.
* For cohort 3 only: Subjects treated with oral Clozapine.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-03 (Estimated)

PRIMARY OUTCOMES:
Safety, rate of adverse events (AEs) | Through study completion, up to 22 weeks for each subject in the first 2 cohorts and up to 24 weeks for each subject in the 3rd cohort
Plasma concentration of cariprazine and its active metabolites (DCAR, DDCAR) | Through study completion, up to 22 weeks for each subject in the first 2 cohorts and up to 24 weeks for each subject in the 3rd cohort

SECONDARY OUTCOMES:
Tolerability - Incidence and severity of injection site reactions | Through study completion, up to 22 weeks for each subject in the first 2 cohorts and up to 24 weeks for each subject in the 3rd cohort
Efficacy - Cohort 3: Positive and Negative Symptom Score (PANSS) | Through study completion, up to 24 weeks for each subject in the 3rd cohort
Efficacy - Cohort 3: Clinical Global Impression Scale (CGI) | Through study completion, up to 24 weeks for each subject in the 3rd cohort

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Clinical Research Center, Ness Ziona
  - Israeli Medical Center for Alzheimer, Ramat Gan
  - Tel Aviv, Israel, Tel Aviv

IPD SHARING:
Plan to Share IPD: No